CLINICAL TRIAL: NCT03385837
Title: Activity Level and Barriers to Participate of Cardiac Rehabilitation in Advanced Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Luciana Diniz Nagem Janot Matos, PhD, Hospital Israelita Albert Einstein
Other Study IDs: 2249-14
Record Dates: First submitted 2017-11-30; First posted 2017-12-29 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure，Congestive; Cardiac Rehabilitation; Physical Exercise
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure Patients: Cardiac Rehabilitation in Advanced Heart Failure Patients

SUMMARY:
A prospective longitudinal and observational clinical study will be conducted with hospitalized heart failure patients.The main purpose is to know the level of physical activity of these patients after their discharge in relation to the orientation received during their hospitalization and identify the barriers perceived by these patients to participate in a cardiac rehabilitation program. The outcomes are available by telephone calls in 30 and 90 days after discharge.

DETAILED DESCRIPTION:
Heart failure is a progression epidemic problem, parallel to population aging. The costs of this disease are estimates in 38 billion of dollars per year, many of those have a relationship to high number of hospitalizations and decompensated heart failure. Non-adherence to drug treatment and non-pharmacological measures as cardiac rehabilitation are the major causes of high number of mortality and hospitalizations by heart failure. Our objectives will be to identify in decompensated heart failure inpatients the level of physical activity that they done before hospitalization, the barriers for the non-use of cardiac rehabilitation and their disposition to changes of lifestyle. Correlation between level of physical activity and readmission in 30 and 90 days after hospital discharge will be done. To understand the profile of these patients and difficulties for to do physical exercise could help to make future actions with focus in to obtain high adherence to changes in lifestyle.

ELIGIBILITY:
Inclusion criteria Patients in the heart failure protocol of the cardiology program with medical release in the next 72 hours

Exclusion criteria

* Inpatients for more than 30 days
* Younger than 18 years old
* Patients not recommended to do exercises (patients with osteoarticular alterations that doesn't allow the performance of physical exercise)
* Patients with cognitive impairment (Mini Mental <24), visual or psychiatric impairment which restrain the comprehension of the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Protocol of heart failure patients will be maped since their hospitalizaztion, however, their approach to get in the study will be fulfilled when they had medical release in 72 hours.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Know the physical activity level in heart failure patients before hospitalization | Before hospitalization
  - To know the physical activity level in heart failure patients before the hospitalization using one questionnaire: the International Physical Activity Questionnaires (IPAQ).
Know cardiac rehabilitation barriers in heart failure patients | At screening
  -To identify the cardiac rehabilitation barriers in heart failure patients using a likert scale CRBS (Cardiac Rehabilitation Barriers Scale) which assesses patients' perceptions regarding the personal (patient), professional (health professional) and institutional (system) barriers that affect participation and adherence to cardiac rehabilitation programs.
Know disposition for changes in life habits | At screening
  - To identify the disposition for changes in life habits related to physical activity using the Disposition Scale described for Prochaska Jo and Diclemente with the results: pre contemplation, contemplation, preparation and action.

SECONDARY OUTCOMES:
Know the change from baseline physical activity level to 30 days after discharge | 30 days
  To know the physical activity level in heart failure patients 30 days after discharge using one questionnaire: the International Physical Activity Questionnaires (IPAQ).
Know the change from baseline physical activity level to 90 days after discharge | 90 days
  To know the physical activity level in heart failure patients 90 days after discharge using one questionnaire: the International Physical Activity Questionnaires (IPAQ).
Adhesion of orientation | 90 days
  Verify the adhesion of the orientation given in the hospitalization about medications and daily weight measure
New hospitalizations 30 and 90 days after discharge | 30 and 90 days
  Verify if there were new hospitalizations and its reasons in this period
Correlate new hospitalization with physical activity and orientations | 90 days
  Correlate the new hospitalization in 30 and 90 days after discharge with the participation in physical activity program and orientation given in the hospital (medications and daily weight measure) in the statistical analysis
Measure anxiety and depression | At screening
  Measure anxiety and depression through HADS (Hospital Anxiety and Depression Scale) which shows if it is impossible, possible or probable.
Measure cognitive impairment | At screening
  Measure if the patient presents cognitive impairment applying the MMSE (Mini-mental State Examination).
Correlate anxiety and depression with cognitive impairment | At screening
  Correlate anxiety and depression with cognitive impairment in the statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Matos, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein 's (IIEP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: ICF
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data acess requests will be reviewed by and internal or external Independent Review Panel. Requestors will be required to sign a Data Acess Agreement.

REFERENCES:
- [Background] Hallal PC, Simoes E, Reichert FF, Azevedo MR, Ramos LR, Pratt M, Brownson RC. Validity and reliability of the telephone-administered international physical activity questionnaire in Brazil. J Phys Act Health. 2010 May;7(3):402-9. doi: 10.1123/jpah.7.3.402. PMID 20551498
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bocchi EA, Braga FG, Ferreira SM, Rohde LE, Oliveira WA, Almeida DR, Moreira Mda C, Bestetti RB, Bordignon S, Azevedo C, Tinoco EM, Rocha RM, Issa VS, Ferraz A, Cruz Fd, Guimaraes GV, Montera Vdos S, Albuquerque DC, Bacal F, Souza GE, Rossi Neto JM, Clausell NO, Martins SM, Siciliano A, Souza Neto JD, Moreira LF, Teixeira RA, Moura LZ, Beck-da-Silva L, Rassi S, Azeka E, Horowitz E, Ramires F, Simoes MV, Castro RB, Salemi VM, Villacorta Junior H, Vila JH, Simoes R, Albanesi F, Montera MW; Sociedasde Brasileira de Cardiologia. [III Brazilian Guidelines on Chronic Heart Failure]. Arq Bras Cardiol. 2009;93(1 Suppl 1):3-70. No abstract available. Portuguese. PMID 20963312
- [Background] Mendes M. Barriers to participation in cardiac rehabilitation programs. Rev Port Cardiol. 2011 May;30(5):509-14. No abstract available. English, Portuguese. PMID 21800479
- [Background] Cabral-de-Oliveira AC, Ramos PS, Araujo CG. Distance from home to exercise site did not influence the adherence of 796 participants. Arq Bras Cardiol. 2012 Jun;98(6):553-8. doi: 10.1590/s0066-782x2012005000039. Epub 2012 Apr 19. English, Portuguese. PMID 22522721
- [Background] Ghisi GL, Santos RZ, Schveitzer V, Barros AL, Recchia TL, Oh P, Benetti M, Grace SL. Development and validation of the Brazilian Portuguese version of the Cardiac Rehabilitation Barriers Scale. Arq Bras Cardiol. 2012 Apr;98(4):344-51. doi: 10.1590/s0066-782x2012005000025. Epub 2012 Mar 15. English, Portuguese. PMID 22426990
- [Result] Mangini S, Pires PV, Braga FG, Bacal F. Decompensated heart failure. Einstein (Sao Paulo). 2013 Jul-Sep;11(3):383-91. doi: 10.1590/s1679-45082013000300022. PMID 24136770
- [Result] Mair V, Breda AP, Nunes ME, Matos LD. Evaluating compliance to a cardiac rehabilitation program in a private general hospital. Einstein (Sao Paulo). 2013 Jul-Sep;11(3):278-84. doi: 10.1590/s1679-45082013000300004. PMID 24136752
- [Result] Rabelo ER, Aliti GB, Goldraich L, Domingues FB, Clausell N, Rohde LE. Non-pharmacological management of patients hospitalized with heart failure at a teaching hospital. Arq Bras Cardiol. 2006 Sep;87(3):352-8. doi: 10.1590/s0066-782x2006001600019. English, Portuguese. PMID 17057937
- [Derived] Carvalho ACSM, Groehs RV, Pereira C, Soares VL, Mota TP, Grace SL, Matos LDNJ. Barriers to cardiac rehabilitation and their association with hospital readmission in patients with heart failure. Einstein (Sao Paulo). 2025 Mar 17;23:eAO0713. doi: 10.31744/einstein_journal/2025AO0713. eCollection 2025. PMID 40105570